CLINICAL TRIAL: NCT02178956
Title: A Phase III Clinical Trial of BBI608 Plus Weekly Paclitaxel vs. Placebo Plus Weekly Paclitaxel in Adult Patients With Advanced, Previously Treated Gastric and Gastro-Esophageal Junction Adenocarcinoma
Brief Title: A Study of BBI608 Plus Weekly Paclitaxel to Treat Gastric and Gastro-Esophageal Junction Cancer
Acronym: BRIGHTER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBI608-336; 2014-000774-18 (EudraCT Number)
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Results first posted 2021-05-10 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — napabucasin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BBI608 plus Paclitaxel (Experimental)
  Interventions: Drug: BBI608; Drug: Paclitaxel
- Placebo plus Paclitaxel (Placebo Comparator)
  Interventions: Drug: Paclitaxel; Other: Placebo

INTERVENTIONS:
Drug: BBI608 — BBI608 480 mg orally two times daily (960 mg total daily dose)
  Other Names: Napabucasin; BB608; BBI-608
  Arms: BBI608 plus Paclitaxel
Drug: Paclitaxel — Paclitaxel 80 mg/m2 I.V. infusion on Days 1, 8, and 15 of every 4-week cycle
Other: Placebo — Orally two times daily
  Arms: Placebo plus Paclitaxel

SUMMARY:
The purpose of this study is to find out whether it is better to receive a new drug, BBI608, in addition to paclitaxel chemotherapy or better to receive paclitaxel chemotherapy alone as second line treatment for gastric and gastroesophageal junction cancer after prior first line platinum and fluoropyrimidine based chemotherapy.

DETAILED DESCRIPTION:
The goal of this study is to determine if paclitaxel given together with BBI608 as second line therapy will prolong overall survival compared to paclitaxel alone.

Approximately 700 patients will be randomized with histologically or cytologically confirmed metastatic gastric or gastroesophageal junction adenocarcinoma.

Patients must have failed first line therapy with any platinum/fluoropyrimidine doublet.

BBI608/placebo will be administered daily, paclitaxel will be administered i.v. on days 1, 8 and 15 of a 4 weekly cycle.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically confirmed advanced gastric or GEJ adenocarcinoma that is metastatic or locally advanced and unresectable.
* Failed treatment with one regimen containing at least a platinum/fluoropyrimidine doublet for unresectable or metastatic disease.Treatment failure is defined as progression of disease (clinical or radiologic) during first line treatment for unresectable or metastatic disease or ≤ 6 months after last dose of first line treatment.
* Paclitaxel therapy is appropriate for the patient and is recommended by the Investigator.
* Imaging investigations including CT/MRI of chest/abdomen/pelvis or other scans as necessary to document all sites of disease done within 21 days prior to randomization. Patients with either measurable disease OR non-measurable evaluable disease will be eligible.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.

  ･≥ 18 years of age.
* For male or female patient of child producing potential: Must agree to use contraception or take measures to avoid pregnancy during the study and for 6 months after the final dose of Paclitaxel or for 30 days for female patients and for 90 days for male patients, of the final BBI608/Placebo dose if Paclitaxel was not administered.
* Women of child bearing potential (WOCBP) must have a negative serum or urine pregnancy test within 5 days prior to randomization.
* Alanine transaminase (ALT) ≤ 3 × institutional upper limit of normal (ULN) [≤ 5 × ULN in presence of liver metastases] within 14 days prior to randomization.
* Hemoglobin (Hgb) ≥ 9.0 g/dL within 14 days prior to randomization. Must not have required transfusion within 1 week of baseline Hgb assessment.
* Total bilirubin ≤ 1.5 × institutional ULN [≤ 2.0 x ULN in presence of liver metastases] within 14 days prior to randomization.
* Creatinine ≤ 1.5 × institutional ULN or Creatinine Clearance > 50 ml/min (as calculated by the Cockroft-Gault equation) within 14 days prior to randomization.
* Absolute neutrophil count ≥ 1.5 x 10^9/L within 14 days prior to randomization.
* Platelet count ≥ 100 x 10^9/L within 14 days prior to randomization. Must not have required transfusion within 1 week of baseline platelet assessment.
* Other baseline laboratory evaluations must be done within 14 days prior to randomization.
* Patient must consent to provision of a representative formalin fixed paraffin block of tumor tissue, if available, in order that the specific correlative marker assays may be conducted.
* Patient must consent to provision of a sample of blood in order that the specific correlative marker assays may be conducted.
* Patients must be accessible for treatment and follow up.
* Protocol treatment is to begin within 2 working days of patient randomization.
* The patient is not receiving therapy in a concurrent clinical study and the patient agrees not to participate in other interventional clinical studies during their participation in this trial while on study treatment. Patients participating in surveys or observational studies are eligible to participate in this study.

Exclusion Criteria:

* Anti-cancer chemotherapy or biologic therapy if administered prior to the first planned dose of BBI608/placebo within period of time equivalent to the usual cycle length of the regimen. An exception is made for oral fluoropyrimidines (e.g. capecitabine, S-1), where a minimum of 10 days since last dose must be observed prior to the first planned dose of BBI608/placebo.Radiotherapy, immunotherapy, or investigational agents within four weeks of first planned dose of BBI608/placebo, with the exception of a single dose of radiation up to 8 Gray (equal to 800 RAD) with palliative intent for pain control up to 14 days before randomization.
* Prior taxanes in the neoadjuvant or adjuvant setting with progression occurring within 6 months of completion of taxane therapy; or any taxanes in the metastatic setting.
* More than one prior chemotherapy regimen administered in the metastatic setting.
* Major surgery within 4 weeks prior to randomization.
* Any known symptomatic brain metastases requiring steroids.
* Women who are pregnant or breastfeeding.
* Gastrointestinal disorder(s) which, in the opinion of the Qualified/Principal Investigator, would significantly impede the absorption of an oral agent.
* Unable or unwilling to swallow BBI608/placebo capsules daily.
* Uncontrolled intercurrent illness.
* Peripheral neuropathy ≥ CTCAE Grade 2 at baseline.
* History of other malignancies except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥ 3 years.
* Prior treatment with BBI608.
* Any active disease condition which would render the protocol treatment dangerous or impair the ability of the patient to receive protocol therapy.
* Any condition (e.g. psychological, geographical, etc.) that does not permit compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 714 (Actual)
Dates: Start 2014-10; Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (262):
- United States (26):
  - Mayo Clinic - Arizona, Scottsdale, Arizona
  - Colorado Cancer Research Program, Denver, Colorado
  - Indiana University Health Goshen Center For Cancer Care, Goshen, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Cancer Center of Kansas, Wichita, Kansas
  - Ochsner NCI CORP, New Orleans, Louisiana
  - Spectrum Health Butterworth, Grand Rapids, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Metro-Minnesota NCI CORP, Saint Louis Park, Minnesota
  - Heartland NCORP, St Louis, Missouri
  - New Hampshire Oncology Hematology - Concord, Concord, New Hampshire
  - New Hampshire Oncology Hematology - Laconia, Laconia, New Hampshire
  - Weill Medical College of Cornell University, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Indiana University Health University Hospital, Chapel Hill, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - The University of Oklahoma Health Sciences Center (OUHSC), Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Cancer Institute/ Swedish Health Services, Seattle, Washington
  - Saint Vincent Hospital CCOP, Green Bay, Wisconsin
  - St. Mary's Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield CCOP, Marshfield, Wisconsin
- Australia (25):
  - Bankstown-Lidcombe, Bankstown, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Central coast area health (public), Gosford, New South Wales
  - Port Macquaries Base Hospital, Port Macquarie, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Riverina Cancer Care Centre, Wagga Wagga, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Sunshine Coast Hospital and Health Service, Nambour, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Bendigo Hospital, Bendigo, Victoria
  - Monash Health, East Bentleigh, Victoria
  - Peninsula & South Eastern Haematology and Oncology Group, East Bentleigh, Victoria
  - St Vincent's Hospital, Fitzroy, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Ballarat base hospital, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - Ballarat Oncology and Haematology Services, Wendouree, Victoria
  - Fiona Stanley Hospital, Subiaco, Western Australia
- Belgium (9):
  - Imelda Ziekenhuis, Bonheiden, Antwerpen
  - UZ Antwerpen, Edegem, Antwerpen
  - Institut Jules Bordet, Brussels, Brussels Capital
  - UZ Brussel - Campus Jette, Brussels, Brussels Capital
  - Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital
  - CHU Ambroise Paré, Mons, Hainaut
  - UZ Leuven - Campus Gasthuisberg, Leuven, Vlaams Brabant
  - AZ Sint-Lucas - Campus Sint-Lucas, Brugge (Assebroek)
  - CHU de Liège - Domaine Universitaire du Sart Tilman, Liège
- Brazil (13):
  - Instituto do Câncer do Ceará - Instituto do Câncer do Cear, Fortaleza, Ceará
  - Oncovida - Centro de Oncologia da Bahia, Salvador, Estado de Bahia
  - Cetus Hospital Dia Oncologia, Belo Horizonte, Minas Gerais
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - Hospital da Cidade de Passo Fundo, Passo Fundo, Rio Grande do Sul
  - UPCO - Unidade de Pesquisa Clinica em Oncologia LTDA, Pelotas, Rio Grande do Sul
  - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Fundaçao dr Amaral Carvalho, Jaú, São Paulo
  - Hospital de Base de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Inca-RJ, Rio de Janeiro
  - IEP São Lucas, São Paulo
  - Casa de Saúde Santa Marcelina, São Paulo
- Bulgaria (7):
  - Specialised Hospital for Active Treatment in Oncology, Sofia, Sofia-Grad
  - UMHAT ""Dr. Georgi Stranski"" Dept. Medical Oncology, Pleven
  - District Dispensery with Stationary - Sofia District, Sofia
  - Multiprofile hospital for active treatment, Sofia
  - UMHAT"Sv.Ivan Rilski", Sofia
  - Uni. Multiprofile Hospital for Active treatment Sveta Marina, Varna
  - COC - Vratsa Dept. of Palliative Care, Vratsa
- Canada (6):
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Saint Michael's Hospital Li Ka Shing Knowledge Institute, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - McGill University Health Centre - Montreal General Hospital, Montreal, Quebec
- China (26):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The 307th Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Southern Medical University, Nanfang Hospital, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Heilongjiang, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The 81 Hospital of the Chinese People's Liberation Army, Nanjing, Jiangsu
  - Jiang Su Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Jilin Cancer Hospital, Jilin, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Xin Jiang Tumor Hospital, Xin Jiang Medical University, Ürümqi, Xinjiang
  - Sir Run Run Shaw Hospital School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Tongji Hospital, Wuhan
- Czechia (5):
  - FN Hradec Kralove, Hradec Králové, Královéhradecký kraj
  - Fakultni nemocnice Olomouc, Olomouc, Olomoucký kraj
  - Masarykuv onkologicky ustav, Brno
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Nemocnice Na Bulovce, Prague
- Estonia (2):
  - East Tallinn Central Hospital Oncology Center, Tallinn, Harju
  - Tartu University Hospital Clinic of Hematology and Oncology, Tartu, Tartu
- France (15):
  - Centre Antoine Lacassagne, Nice, Alpes-Maritimes
  - Hopital Saint Joseph - Marseille, Marseille, Bouches-du-Rhône
  - Centre Paul Papin, Saint-Herblain, Loire-Atlantique
  - Centre Rene Gauducheau, Saint-Herblain, Loire-Atlantique
  - Hopital Privé Jean Mermoz, Lyon, Rhône
  - Chd Vendee La Roche Sur Yon, La Roche-sur-Yon, Vendée
  - Hospital of Poitiers, Poitiers, Vienne
  - Hôpital Morvan - CHRU de Brest, Brest
  - CHU Estaing, Clermont-Ferrand
  - CHU - Hôpital De La Timone, Marseille
  - Centre Hospitalier De Mont De Marsan - Hopital Layné, Mont-de-Marsan
  - Centre eugène marquis, Rennes
  - CHU Saint Etienne, Saint-Etienne
  - Centre Hospitalier Universitaire (CHU) de Toulouse - Hopital, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (12):
  - Klinikum Bogenhausen, München, Bavaria
  - Klinikum der Johann Wolfgang Goethe-Universität, Frankfurt am Main, Hesse
  - Ev. Krankenhaus Bielefeld, Bielefeld, North Rhine-Westphalia
  - Kliniken Essen-Mitte Evang. Huyssens-Stiftung, Essen, North Rhine-Westphalia
  - Johannes Gutenberg-Universitaet, Maintz, Rhineland-Palatinate
  - Universitätsklinik Carl-Gustav-Carus Dresden, Dresden, Saxony
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Charite - Campus Benjamin Franklin (Cbf), Berlin
  - Charite, Berlin
  - Klinikum Esslingen, Esslingen am Neckar
  - Facharztzentrum Eppendorf, Hamburg
  - OncoResearch Lerchenfeld GmbH, Hamburg
- Hungary (10):
  - Pécsi Tudományegyetem Klinikai Központ, Pécs, Baranya
  - Békés Megyei Pándy Kálmán Kórház, Gyula, Bekes County
  - Petz Aladár Megyei Oktató Kórház, Győr, Győr-Moson-Sopron
  - Debreceni Egyetem Klinikai Központ, Debrecen, Hajdú-Bihar
  - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház- Rendelőinté, Szolnok, Jász-Nagykun-Szolnok
  - Josa Andras Oktato Korhaza, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Semmelweis Egyetem, Budapest
  - Egyesített Szent István és Szent László Kórház-Rendelőintéze, Budapest
  - Országos Onkológiai Intézet, Budapest
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
- Israel (7):
  - The E. Wolfson Medical Center [Oncology], Holon, Central District
  - Meir Medical Center, Kfar Saba, Central District
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva, Central District
  - Hadassah Medical Organisation, Jerusalem, Jerusalem
  - Soroka Medical Center [Oncology], Beersheba, Southern District
  - Tel Aviv Sourasky Medical Center, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus, Haifa
- Italy (14):
  - Irccs Irst, Meldola, Forli
  - AUSL della Romagna, Osp. degli Infermi, Faenza, Ravenna
  - Ospedale Umberto I, AOU Ospedali Riuniti Umberto I - GM.Lanc, Ancona
  - IRCCS Ospedale Oncologico "Giovanni Paolo II", Bari
  - Humanitas Gavazzeni, Bergamo
  - Policlinico S.Orsola Malpighi, AOU di Bologna, Bologna
  - PO Garibaldi-Nesima, ARNAS Garibaldi, Catania
  - Azienda Ospedaliera "Istituti Ospitalieri" di Cremona, Cremona
  - AOU S.Martino, IRCCS, IST-Istituto Nazionale Ricerca Sul Can, Genova
  - Azienda Ospedaliera Fatebenefratelli e Oftalmico, Milan
  - Istituto Oncologico Veneto IOV-IRCCS, Padua
  - Ospedale Guglielmo da Saliceto, AUSL Piacenza, Piacenza
  - Unità di Biostatistica e Sperimentazioni Cliniche IRST, Ravenna
  - Ospedale Molinette, AO Città della Salute e della Scienza di, Torino
- Japan (15):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Saku Central Hospital Advanced Care Center, Saku, Nagano
  - Osaka University Hospital, Suita, Osaka
  - Saitama Cancer Center, Kita-Adachi, Saitama
  - Shizuoka Cancer Center, Sunto, Shizuoka
  - Tochigi Cancer Center, Utsunomiya, Tochigi
  - National Cancer Center Hospital, Chūō, Tokyo
  - Kyorin University Hospial, Mitaka, Tokyo
  - Chiba Cancer Center, Chiba
  - Gifu University Hospital, Gifu
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka
- Lithuania (7):
  - Hospital of Lithuanian University of Health sciences, Kaunas, Kaunas County
  - Hospital of Lithuanian University of Health Sciences, Kaunas, Kaunas County
  - Respublikine Panevezio ligonine, Panevezys, Panevežio Apskritis
  - National Cancer Institute, Vilnius, Vilnius County
  - Klaipeda University Hospital, Klaipėda
  - Vilniaus Universiteto ligonines Santariskiu Klinikos, Vilnius
  - Siauliai County Hospital, Šiauliai, Šiauliu Apskritis
- Poland (10):
  - NZOZ Centrum Medyczne HCP Lecznictwo Stacjonarne, Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im. F.Lukaszczyka, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Szpital Specjalistyczny im. L. Rydygiera w Krakowie, Krakow, Lesser Poland Voivodeship
  - Europejskie Centrum Zdrowia Otwock, Szpital im. F. Chopina, Otwock, Masovian Voivodeship
  - Centrum Onkologii Instytut im. M. Sklodowskiej-Curie, Warsaw, Masovian Voivodeship
  - Magodent sp. z o.o. Szpital Onkologiczny, Warsaw, Masovian Voivodeship
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Ośrodek Onko, Brzozów, Podkarpackie Voivodeship
  - Wojewodzkie Centrum Onkologii w Gdansku, Gdansk, Pomeranian Voivodeship
  - Zachodniopomorskie Centrum Onkologii, Szczecin, West Pomeranian Voivodeship
  - Wojewodzki Szpital Specjalistyczny im. M.Kopernika, Lodz, Łódź Voivodeship
- Romania (12):
  - Radiotherapy Center CJ radioterapie si chimioterapie adulti, Floreşti, Cluj
  - Centrul de Oncologie Sf. Nectarie, Craiova, Dolj
  - Oncolab, Craiova, Dolj
  - Institutul Regional de Oncologie Iasi, Lasi, Lasi
  - Sp. Jud. de Urg. "Dr. Constantin Opris" Baia Mare, Baia Mare, Maramureş
  - Oncomed, Timișoara, Timiș County
  - Spitalul Clinic Municipal de Urgenta Timisoara, Timișoara, Timiș County
  - Med Life, Bucharest
  - Spitalul Clinic CF 2, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Centrul de Oncologie Euroclinic, Iași
  - Spitalul Clinic Judetean de Urgenta Sibiu, Sibiu
- Russia (11):
  - Republican Clinical Oncology Dispensary, Ufa, Bahkortostan, Respublika
  - Military Medical Academy n.a. S.M. Kirov, Saint Petersburg, Leningradskaya Oblast'
  - Russian Oncological Research Center n.a. N.N. Blokhin RAMS, Moscow, Moscow
  - City Clinical Hospital #40, Moscow, Moscow
  - GUZ Perm Regional Oncology Dispensary, Perm, Permskiy Kray
  - Northwestern State Medical University n.a. Mechnikov, Saint Petersburg, Sankt-Peterburg
  - First Pavlov State Medical University of Saint-Petersburg, Saint Petersburg, Sankt-Peterburg
  - GBUZ Saint Petersburg clinical scientific and practical cent, Saint Petersburg, Sankt-Peterburg
  - SPb State Budget Institution Oncology Dispansery, Saint Petersburg, Sankt-Peterburg
  - GBUZ of Stavropol Territory Pyatigorsk Oncology Dispensary, Pyatigorsk, Stavropol Kray
  - Guz Clinical Oncology Dispensary #1, Krasnodar
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam, Gyeonggido
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi
  - Asan medical Center, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
- Spain (17):
  - H.U.V. Macarena, Seville, Andalusia
  - Institut Català d'Oncologia-Hospital Germans Trias i Pujol, Badalona, Barcelona
  - C.A.AV-H.Ntra.Sra.de Sonsoles, Ávila, Castille and León
  - H.U.P Hierro-Majadahonda, Majadahonda, Madrid
  - H.del Mar, Barcelona
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - H.Sta.Creu i St.Pau, Barcelona
  - H.U. de Burgos, Burgos
  - Institut Catalá d´Oncología (I.C.O.), L'Hospitalet de Llobregat
  - H.G.U. G. Marañón, Madrid
  - M.D. Anderson Cancer Center Madrid, Madrid
  - H.U. R. y Cajal, Madrid
  - H.C. S.Carlos, Madrid
  - H.U.V.Arrixaca, Murcia
  - H.U.V. del Rocío, Seville
  - C.H.G.U.de Valencia, Valencia
  - H.U. Miguel Servet, Zaragoza
- United Kingdom (9):
  - Aberdeen Royal Infirmary, Aberdeen, Aberdeen City
  - The Beatson West Of Scotland Cancer Centre, Glasgow, Glasgow City
  - Royal Surrey County Hospital, Guildford, Surrey
  - The Royal Marsden Hospital, Sutton, Surrey
  - The Royal Marsden NHS Foundation Trust - Royal Marsden Hospital, Sutton, Surrey
  - Belfast City Hospital, Belfast
  - St. Georges Hospital, London
  - Christie Hospital NHS Foundation Trust, Manchester
  - Southampton University Hospital, Southampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 714 patients were enrolled to this study from 02OCT2014 to 20SEP2017 across 204 sites in 22 countries.
Pre-assignment Details: Study arm was determined at patient randomization to the study, no pre-assignment activities occurred.
Groups:
- Napabucasin + Paclitaxel: Napabucasin was administered orally, twice daily, with doses separated by 12 hours. Paclitaxel 80 mg/m2 (intravenous [IV]) was administered weekly, on Days 1, 8, and 15 of each 28 day study cycle. Napabucasin administration began 2 days prior to the first paclitaxel infusion in the initial run in period.
- Placebo + Paclitaxel: Placebo was administered orally, twice daily, with doses separated by 12 hours. Paclitaxel 80 mg/m2 (intravenous [IV]) was administered weekly, on Days 1, 8, and 15 of each 28 day study cycle. Placebo administration began 2 days prior to the first paclitaxel infusion in the initial run in period.
Period: Overall Study
Arm/Group | Napabucasin + Paclitaxel | Placebo + Paclitaxel
Started | 357 | 357
Completed | 286 | 279
Not Completed | 71 | 78
Not completed — Lost to Follow-up | 4 | 4
Not completed — Sponsor terminated study | 49 | 58
Not completed — Withdrawal by Subject | 15 | 11
Not completed — Various Reasons | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Napabucasin + Paclitaxel | Placebo + Paclitaxel | Total
Number analyzed (Participants) | 357 | 357 | 714
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.787 (11.5130) | 59.887 (11.1231) | 60.337 (11.3207)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 103 | 199
  Male | 261 | 254 | 515
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 107 | 102 | 209
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 237 | 240 | 477
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 11 | 22
ECOG [Count of Participants; unit: Participants] — The ECOG Performance Status describes a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.). The higher the score, the more restricted the patient is clinically determined to be.
  Participants
    0: Fully active, able to carry on all pre-disease performance without restriction | 128 | 134 | 262
    1: Restricted in physically strenuous activity but ambulatory, can carry out light/sedentary work | 229 | 223 | 452
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.24 (4.481) | 23.56 (4.709) | 23.40 (4.596)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: The primary objective of this study is to assess the effect of orally administered BBI608 plus weekly paclitaxel, in comparison to placebo plus weekly paclitaxel on the Overall Survival of patients with advanced histopathologically confirmed gastric or gastroesophageal junction adenocarcinoma who failed treatment with one platinum/fluoropyrimidine containing regimen for unresectable or metastatic disease.
Time Frame: 36 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Napabucasin + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 357 | 357
Months | 6.93 [6.28 to 7.69] | 7.36 [6.64 to 8.15]
Statistical Analysis 1: Comparison: Napabucasin + Paclitaxel vs Placebo + Paclitaxel; Test type: Superiority; p = 0.8596, Log Rank — two-sided; stratified log rank test stratified by region, time to progression on 1st line therapy and disease measurability; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.86 to 1.02] — HR is for napabucasin + Paclitaxel vs Placebo + Paclitaxel. Based on Cox Proportional hazards model stratified by actual stratification variables including region, time to progression on first line therapy and disease measurability

2. Secondary Outcome: Progression Free Survival
Description: Defined as the time from randomization to the first objective documentation of disease progression or death due to any cause which comes first. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria(RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in anon-target lesion, or the appearance of new lesions.
Time Frame: 36 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Napabucasin + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 357 | 357
Months | 3.55 [3.22 to 3.68] | 3.68 [3.48 to 3.71]
Statistical Analysis 1: Comparison: Napabucasin + Paclitaxel vs Placebo + Paclitaxel; Test type: Superiority; p = 0.9028, Log Rank — two sided; stratified log rank test stratified by region, time to progression on 1st line therapy and disease measurability; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.85 to 1.19] — HR is for napabucuasin + Paclitaxel vs Placebo + Paclitaxel. Based on Cox Proportional hazards model stratified by actual stratification variables including region, time to progression on first line therapy and disease measurability

3. Secondary Outcome: Objective Response Rate
Description: Objective Response Rate is defined as the percentage of patients with a documented complete response or partial response (CR + PR) based on RECIST 1.1.
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Groups:
- Napabucasin + Paclitaxel: Napabucasin was administered orally, twice daily, with doses separated by 12 hours. Paclitaxel 80 mg/m2 (intravenous [IV]) was administered weekly, on Days 1, 8, and 15 of each 28 day study cycle. Napabucasin administration began 2 days prior to the first paclitaxel infusion in the initial run in period. Patients were included in this group had a baseline scan and at least one assessment a minimum of 6 weeks from baseline.
- Placebo + Paclitaxel: Placebo was administered orally, twice daily, with doses separated by 12 hours. Paclitaxel 80 mg/m2 (intravenous [IV]) was administered weekly, on Days 1, 8, and 15 of each 28 day study cycle. Placebo administration began 2 days prior to the first paclitaxel infusion in the initial run in period. Patients were included in this group had a baseline scan and at least one assessment a minimum of 6 weeks from baseline.
Arm/Group | Napabucasin + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 289 | 283
Participants | 16 | 18
Statistical Analysis 1: Comparison: Napabucasin + Paclitaxel vs Placebo + Paclitaxel; Test type: Superiority; p = 0.7359, Cochran-Mantel-Haenszel — 2-sided; Based on CMH test stratified by actual stratification variables at baseline including region, and time to progression on first-line therapy; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.60 to 1.44] — Odds ratio for napabucasin vs. Placebo. Based on Logistic Regression Model adjusting for actual Stratification variables at baseline including region, and time to progression on first-line therapy

4. Secondary Outcome: Disease Control Rate
Description: Disease control Rate is defined as the percentage of patients with a documented complete response or partial response (CR + PR+SD) based on RECIST 1.1.
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Napabucasin + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 289 | 283
Participants | 55 | 58
Statistical Analysis 1: Comparison: Napabucasin + Paclitaxel vs Placebo + Paclitaxel; Test type: Superiority; p = 0.6555, Cochran-Mantel-Haenszel — 2-sided; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.66 to 1.30] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Number of Patients With Adverse Events
Description: All patients who have received at least one dose of BBI608/Placebo will be included in the safety analysis. The number of patients who experienced at least one adverse event is reported.
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Groups:
- Napabucasin + Paclitaxel: Napabucasin was administered orally, twice daily, with doses separated by 12 hours. Paclitaxel 80 mg/m2 (intravenous [IV]) was administered weekly, on Days 1, 8, and 15 of each 28 day study cycle. Napabucasin administration began 2 days prior to the first paclitaxel infusion in the initial run in period. Patients included this group received at least one dose of study drug.
- Placebo + Paclitaxel: Placebo was administered orally, twice daily, with doses separated by 12 hours. Paclitaxel 80 mg/m2 (intravenous [IV]) was administered weekly, on Days 1, 8, and 15 of each 28 day study cycle. Placebo administration began 2 days prior to the first paclitaxel infusion in the initial run in period. Patients included this group received at least one dose of study drug.
Arm/Group | Napabucasin + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 357 | 350
Participants | 352 | 338

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time the patient signed informed consent until 30 days after the last protocol treatment administration.
Arm/Group | Napabucasin + Paclitaxel | Placebo + Paclitaxel
All-Cause Mortality (participants affected / at risk) | 286/357 | 275/350
Serious Adverse Events (participants affected / at risk) | 125/357 | 101/350
Other Adverse Events (participants affected / at risk) | 352/357 | 338/350
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Napabucasin + Paclitaxel (N=357) | Placebo + Paclitaxel (N=350)
Vomiting (Gastrointestinal disorders) | 14 | 2
Nausea (Gastrointestinal disorders) | 6 | 0
Abdominal Pain (Gastrointestinal disorders) | 8 | 5
Diarrhoea (Gastrointestinal disorders) | 10 | 3
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 4 | 3
Intestinal obstruction (Gastrointestinal disorders) | 5 | 3
Ascites (Gastrointestinal disorders) | 3 | 3
Dysphagia (Gastrointestinal disorders) | 3 | 5
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 2
Abdominal distension (Gastrointestinal disorders) | 2 | 1
Colitis (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Ileus (Gastrointestinal disorders) | 2 | 3
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 4
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Gastric stenosis (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 3
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Jejunal stenosis (Gastrointestinal disorders) | 1 | 0
Large intestine obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 4
Respiratory tract infection (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 3 | 2
Lung infection (Infections and infestations) | 4 | 3
Peritonitis (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 2 | 1
Septic shock (Infections and infestations) | 2 | 1
Abdominal infection (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 2
Herpes zoster (Infections and infestations) | 1 | 0
Pyonephrosis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Fatigue (General disorders) | 5 | 0
Pyrexia (General disorders) | 6 | 6
Adverse event (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 3 | 1
Asthenia (General disorders) | 4 | 3
Death (General disorders) | 0 | 3
Hyperthermia (General disorders) | 0 | 1
Sudden death (Hepatobiliary disorders) | 1 | 0
Stent malfunction (General disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 2
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Circulatory collapse (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 6 | 5
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Bone marrow (Blood and lymphatic system disorders) | 2 | 0
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 3 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Renal injury (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Bile duct obstruction (Hepatobiliary disorders) | 1 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Napabucasin + Paclitaxel (N=357) | Placebo + Paclitaxel (N=350)
Diarrhoea (Gastrointestinal disorders) | 304 | 126
Nausea (Gastrointestinal disorders) | 178 | 123
Abdominal pain (Gastrointestinal disorders) | 140 | 93
Vomiting (Gastrointestinal disorders) | 135 | 95
Constipation (Gastrointestinal disorders) | 61 | 78
Abdominal pain upper (Gastrointestinal disorders) | 35 | 40
Abdominal distension (Gastrointestinal disorders) | 28 | 25
Dysphagia (Gastrointestinal disorders) | 22 | 24
Ascites (Gastrointestinal disorders) | 18 | 17
Fatigue (General disorders) | 110 | 92
Asthenia (General disorders) | 73 | 73
Pyrexia (General disorders) | 57 | 40
Oedema peripheral (General disorders) | 38 | 31
Decreased appetite (Metabolism and nutrition disorders) | 129 | 103
Hypokalaemia (Metabolism and nutrition disorders) | 29 | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 20 | 18
Neuropathy peripheral (Nervous system disorders) | 46 | 38
Peripheral sensory neuropathy (Nervous system disorders) | 37 | 47
Dysgeusia (Nervous system disorders) | 27 | 15
Dizziness (Nervous system disorders) | 19 | 19
Paraesthesia (Nervous system disorders) | 17 | 22
Anaemia (Blood and lymphatic system disorders) | 126 | 118
Neutropenia (Blood and lymphatic system disorders) | 37 | 49
Leukopenia (Blood and lymphatic system disorders) | 22 | 19
Neutrophil count decreased (Investigations) | 48 | 53
Weight decreased (Investigations) | 41 | 23
White blood cell count decreased (Investigations) | 35 | 43
Alopecia (Skin and subcutaneous tissue disorders) | 73 | 94
Urinary tract infection (Infections and infestations) | 29 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 35 | 34
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 | 37
Chromaturia (Renal and urinary disorders) | 47 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 31 | 33
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 28
Insomnia (Psychiatric disorders) | 30 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT02178956/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT02178956/SAP_001.pdf